CLINICAL TRIAL: NCT02941302
Title: Multimodality Imaging Combined With Multiple Targets Pathological Examination for Detecting of Biological Borders of Gliomas: a Clinical Application Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: xhechun3
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Glioma
Keywords: gliomas; biological boundary; imaging border; operation
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- determine the biological boundaries (Experimental): Neural navigation combined with Intraoperative ultrasound detecting the borders of gliomas, In accordance with established plan to collect multiple targets undergo pathological examination and contrast with imaging boundary to determine the biological boundaries.
  Interventions: Procedure: Detecting of Biological Borders of Gliomas

INTERVENTIONS:
Procedure: Detecting of Biological Borders of Gliomas — Neural navigation combined with Intraoperative ultrasound detecting the borders of gliomas, In accordance with established plan to collect multiple targets undergo pathological examination and contrast with imaging boundary to determine the biological boundaries.

SUMMARY:
Knowledge of the spatial extent of gliomas is an essential prerequisite for the treatment planning. In particular, the localization of the border zone between tumor infiltrated and normal brain tissue is one of the major problems to be solved before beginning therapy. However, it is a well known problem that, in conventional magnetic resonance imaging (MRI), it often is difficult to detect areas with low tumor infiltration, especially in gliomas, because of their infiltrative and often diffuse nature.The study has two purpose:I.To correlate the imaging border zone with pathological grade of different tumor site following surgery in patients with newly diagnosed intracranial gliomas, work out the biological border zone, and complete resect the tumor.II.To determine the feasibility of defining the optimal target volume for radiation therapy using MR spectroscopy, diffusion, perfusion and functional imaging.

DETAILED DESCRIPTION:
Gliomas are widely infiltrative tumors. Although an oncological resection is not feasible, there is compelling evidence that patients benefit from resection of the tumor. The surgical target is the main tumor bulk, which is defined as the contrast enhancing part of the tumor on preoperative MRI. Surgical treatment in gliomas is based on maximal safe resection of this mass. Several new technologies have been devised to maximize the resection and intraoperative MRI is one of these new technologies. Intraoperative MRI has been shown by many studies to increase the extent of resection in glioma surgery. Intraoperative determination of the extent of resection, however, requires use of intravenous contrast administration, which has some technical limitations. Fundamental problems associated with the use of contrast material are the enhancement at the resection margin and contrast leakage into the resection cavity. Both problems can complicate the differential diagnosis between residual tumor and surgically induced changes. Nowadays, the basic theory of a largest removal the tumor is the imaging boundary.

Knowledge of the spatial extent of gliomas is an essential prerequisite for the treatment planning. In particular, the localization of the border zone between tumor infiltrated and normal brain tissue is one of the major problems to be solved before beginning therapy. However, it is a well known problem that, in conventional magnetic resonance imaging (MRI), it often is difficult to detect areas with low tumor infiltration, especially in gliomas, because of their infiltrative and often diffuse nature.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed intracranial glioma
* A diagnostic contrast enhanced CT/MRI demonstrating the lesion prior to registration
* Patient must sign a study specific informed consent form; if the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the patient's legal representative

Exclusion Criteria:

* Patient without brain gliomas
* Inability to obtain histological proof of glioma (functional domain and particular domain)
* Psychiatric conditions precluding informed consent
* Patients who cannot tolerate operation
* Patients who are pregnant or breast feeding
* Urine pregnancy test will be performed on women of child bearing potential

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
the biological border zone of glioma | during the operation
  Neural navigation combined with Intraoperative ultrasound detecting the borders of gliomas, In accordance with established plan to collect multiple targets undergo pathological examination and contrast with imaging boundary to determine the biological boundaries.Pathological specimen collection:Marked by the tumor center, in a clockwise order of the maximum geometric figure of the tumor:1.Front boundary. 2.Right boundary. 3.Rear boundary. 4.Left boundary. 5.Deepest part

SECONDARY OUTCOMES:
the degree of surgical resection of gliomas | 24 hours after operation

OTHER OUTCOMES:
the optimal target volume for radiation therapy | 3 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Xia hechun, M.D., Study Chair — General Hospital of Ningxia Medical University; Wang Xiaodong, M.D., Principal Investigator — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No